CLINICAL TRIAL: NCT00523211
Title: Vicriviroc in Combination Treatment With an Optimized ART Regimen in HIV-Infected Treatment-Experienced Subjects (VICTOR-E3)
Brief Title: Vicriviroc in HIV-Treatment Experienced Subjects (Study P04405AM5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04405; 3553293
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: Acquired Immunodeficiency Syndrome; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Arm (Experimental): Vicriviroc 30 mg QD
  Interventions: Drug: Vicriviroc
- Placebo Control Arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vicriviroc — One tablet of vicriviroc 30 mg once daily.
  Other Names: SCH 417690
  Arms: Test Arm
Drug: Placebo — One tablet of placebo once daily.
  Arms: Placebo Control Arm

SUMMARY:
Vicriviroc (vye-kri-VYE-rock) is an investigational drug (not yet approved by Government Regulatory Authorities for commercial use) that belongs to a new class of drugs, called CCR5 receptor blockers. This group of drugs blocks one of the ways HIV enters T-cells (the cells that fight infection). Previous smaller studies in HIV treatment-experienced patients, have shown that vicriviroc is safe and effective. The purpose of this study is to confirm the previous findings in a larger phase 3 study over a 48-week period, and show that when taken in combination with other appropriate HIV drugs, vicriviroc can decrease the level of HIV (viral load) in the blood and that it is well tolerated.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-center study of vicriviroc maleate in HIV subjects infected with CCR5-tropic virus only and who have documented

resistance to at least 2 of the 3 antiretroviral drug classes (NRTI, NNRTI or PI) or at least 6 months experience with at

least 2 of the following: one NRTI, one NNRTI, or two PIs (excluding low-dose ritonavir)and failed at least one standard triple-drug regimen. The study will compare the virologic benefit of adding vicriviroc to an optimized background regimen to a control group receiving placebo plus the new optimized background therapy. The optimized background regimen will be chosen by the investigator based on results of drug susceptibility tests performed at Screening, history of prior antiretroviral drug use by the patient, and drug toxicity. OBT must include a PI boosted by ritonavir (>=100 mg ritonavir), and at least 2 active drugs (ie, to which HIV isolate is fully susceptible). Primary efficacy analysis will be conducted when all subjects have completed 48 weeks of treatment. An interim analysis will be performed when all subjects have completed 24 weeks of treatment. After completing Week 48 of the study, subjects who meet applicable criteria will be offered open-label vicriviroc 30 mg QD, if appropriate until the sponsor terminates the clinical development of vicriviroc. Additionally, subjects who discontinued early from the study prior to Week 48 may be eligible for the open-label segment of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be infected with HIV-1 virus.
* Subject must have documented plasma HIV-1 RNA >1000 copies/mL within 60 days of Visit 1/Day 1 (randomization) and must be either

  * on a stable regimen of 3 or more antiretrovirals (ART) for at least 4

weeks prior to the screening visit

OR

* on no ART agents for at least 4 weeks prior to

the screening visit.

* Subject must be ART experienced and have documented resistance to at least 2 of the following 3 drug classes: nucleoside reverse transcriptase inhibitor (NRTI); non-nucleoside reverse transcriptase inhibitor (NNRTI); or protease inhibitor (PI)

OR

Subject must have ART class experience for at least 6 months with at least two of the following: one NRTI; one NNRTI; two PIs (excluding low-dose ritonavir).

* Women of child-bearing potential must agree to use a medically accepted method of contraceptive as defined by the protocol.
* Subject must be willing to initiate CD4+ cell count-guided chemoprophylaxis to prevent opportunistic infection as defined in protocol.

Exclusion Criteria:

* Subjects with detectable CXCR4-tropic or dual/mixed CCR5/CXCR4-tropic HIV isolates at Screening.
* Subjects with prior history of malignancy (with exceptions of cutaneous Kaposi's sarcoma without visceral or mucosal involvement that resolved with HAART but without systemic anti-cancer treatment, and basal-cell carcinoma of skin); or prior receipt of cytotoxic cancer chemotherapy that may increase the risk of malignancy.
* Subjects with seizure disorder requiring anti-seizure therapy or with any condition that is likely to increase risk of seizure (CNS malignancy or toxoplasmosis).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with undetectable plasma HIV-1 RNA (<50 copies/mL) | 48 weeks

SECONDARY OUTCOMES:
Mean change from baseline in plasma HIV-1 RNA (log10 copies/mL); Proportion of subjects with <400 copies/mL of plasma HIV-1 RNA; Proportion of subjects with >=2log10 reduction from baseline in plasma HIV-1 RNA | 48 weeks

REFERENCES:
- [Derived] Caseiro MM, Nelson M, Diaz RS, Gathe J, de Andrade Neto JL, Slim J, Solano A, Netto EM, Mak C, Shen J, Greaves W, Dunkle LM, Vilchez RA, Zeinecker J. Vicriviroc plus optimized background therapy for treatment-experienced subjects with CCR5 HIV-1 infection: final results of two randomized phase III trials. J Infect. 2012 Oct;65(4):326-35. doi: 10.1016/j.jinf.2012.05.008. Epub 2012 May 24. PMID 22634184